CLINICAL TRIAL: NCT05141747
Title: An Open-label, Multi-center, Phase II Clinical Study to Evaluate the Safety, Efficacy and Pharmacokinetics of MRG002 in Patients With HER2-positive/HER2-low Locally Advanced or Metastatic Gastric/ Gastroesophageal Junction Cancer.
Brief Title: A Study of MRG002 in the Treatment of HER2-positive/HER2-low Locally Advanced or Metastatic Gastric/Gastroesophageal Junction Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-007
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Locally Advanced Gastric Cancer; Metastatic HER2 Positive Gastroesophageal Junction Cancer
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2; Gastric/Gastroesophageal Junction Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG002 (Experimental): MRG002 will be administrated by an IV infusion of 2.6 mg/kg on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG002 as single agent in patients with HER2-positive /HER2-low locally advanced or metastatic gastric/ gastroesophageal junction cancer.

DETAILED DESCRIPTION:
There are two cohorts in this study. HER2-positive and HER2-low patients will be allocated to cohort 1 and cohort 2, respectively. When the 20th, 40th, or 60th patient in each cohort completed at least one post-baseline tumor assessment, the Safety Monitoring Committee will review the safety and efficacy of these patients to determine dose selection, enrollment continuation, study population, and sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the ICF and follow the requirements specified in the protocol.
2. Aged ≥18.
3. Life expectancy ≥ 3 months.
4. Patients with histologically or cytologically confirmed gastric/ gastroesophageal junction cancer.
5. In Cohort 1, a positive HER2 test result defined as follows: IHC 3+ or IHC 2+ and ISH positive. In Cohort 2, low HER2 expression defined as follows: IHC 1+, or IHC 2+ and ISH negative.
6. Documented tumor progression or intolerance during or after at least one prior line of platinum- and/or fluoropyrimidine-based chemotherapy ± anti-HER2 (trastuzumab or equivalent) therapy.
7. Willing and able to provide adequate archival tumor tissue samples for HER2 status confirmation by central laboratory.
8. Cohort 1 patients, who have received prior anti-HER2 therapy, are willing to undergo fresh tissue biopsy to confirm HER2 status as assessed by the investigator to be feasible and safe.
9. Patients must have at least one measurable tumor lesion according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
10. The score of ECOG for performance status is 0 or 1 with no deterioration within 2 weeks prior to the first dose of the study drug.
11. Organ function must meet the basic requirements.

Exclusion Criteria:

1. Patients with the following pathological diagnosis: squamous cell carcinoma, carcinoid tumor, neuroendocrine carcinoma, undifferentiated carcinoma, or other unclassifiable gastric cancer.
2. Peripheral neuropathy ≥ Grade 2 per CTCAE 5.0.
3. Prior treatment with HER2-targeted ADC.
4. Known allergic reaction to any component or excipient of MRG002, or known allergic reaction to trastuzumab or other prior anti-HER2 or other monoclonal antibodies ≥ Grade 3.
5. Presence of untreated or uncontrolled central nervous system (CNS) metastases.
6. Patients received chemotherapy, biological therapy, radical radiotherapy or other anti-tumor treatment within 3 weeks prior to the first dose of the study drug.
7. Any severe cardiac dysfunction, history of myocardial infarction, stroke, or transient ischemic attack (TIA) within 6 months prior to enrollment.
8. Pulmonary embolism or deep venous thrombosis within 3 months prior to the first dose of the study drug.
9. Tumor lesions with bleeding tendency or treated with blood transfusion within 2 weeks prior to the first dose of the study drug.
10. Toxicities due to prior anti-cancer therapy have not resolved to ≤ Grade 1 (CTCAE v5.0).
11. Concurrent malignancy within 5 years prior to enrollment.
12. Uncontrolled high blood pressure and diabetes.
13. History of ventricular tachycardia or torsades de pointes. Any clinically significant abnormalities in rhythm, conduction, or morphology on the resting ECG.
14. History of moderate to severe dyspnea at rest due to advanced cancer or its complications, severe primary lung disease, current need for continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonitis.
15. Patients who had undergone thoracotomy, laparotomy, or surgery requiring general anesthesia without complete recovery within 4 weeks prior to the first dose of the study drug.
16. Active hepatitis B, active hepatitis C, syphilis or human immunodeficiency virus (HIV) infection.
17. Active uncontrolled bacterial, viral, fungal, rickettsial, or parasitic infection requiring intravenous anti-infective therapy within 2 weeks prior to the first dose of study drug.
18. Any severe and/or uncontrolled systemic diseases.
19. Use of systemic corticosteroids within 4 weeks prior to the first dose of study drug.
20. Use of potent CYP3A4 inhibitors or potent CYP3A4 inducers within 2 weeks prior to the first dose of study drug or need to continue during the study.
21. Female patents with a positive serum pregnancy test or who are breast-feeding or who do not agree to take adequate contraceptive measures during the treatment and for 180 days after the last dose of study treatment.
22. Other conditions inappropriate for participation in this clinical trial, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to study completion, up to 24 months
  ORR is defined as the percentage of patients with a complete response (CR) and partial response (PR) according to RECIST v1.1.
Adverse Events (AEs) | Baseline to 45 days after the lase dose of study treatment.
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Baseline to study completion, up to 24 months.
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion, up to 24 months.
  OS is defined as the duration from the start of treatment to death of any cause.
Duration of Response (DoR) | Baseline to study completion, up to 24 months.
  DOR is defined as the time from first documented objective response to the first onset of tumor progression or death of any cause.
Disease Control Rate (DCR) | Baseline to study completion, up to 24 months.
  DCR is defined as the percentage of patients who achieve CR, PR, and stable disease (SD) after treatment.
Pharmacokinetics (PK) Parameter of MRG002: concentration-time curve | Baseline to 30 days after the last dose of study treatment
  Plot of drug concentration changing with time after drug administration.
Immunogenicity (ADA) | Baseline to 30 days after the last dose of study treatment.
  The proportion of patients with positive ADA results.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Sciences and Peking Union Medical College; Jin Li, MD, Principal Investigator — Shanghai Oriental Hospital
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No